CLINICAL TRIAL: NCT06468254
Title: An Exploratory Clinical Study of Statins for Improving Chemotherapy and Maintenance in Patients With Ovarian Cancer: a Prospective, Multicenter Clinical Study
Brief Title: An Exploratory Clinical Study of Statins for Improving Chemotherapy and Maintenance in Patients With Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Bai-Rong Xia, Chairman of Department of Gynaecology Surgery, Anhui Provincial Cancer Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024 NO. 049
Record Dates: First submitted 2024-05-27; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Ovarian Cancer
Keywords: Statins
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Sugars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Statin Group (Experimental): Statins, 40 mg daily for 1 year or with dosage adjusted based on patient tolerance
  Interventions: Drug: Statin
- Control Group (Placebo Comparator): Sugar pill daily for 1 year
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Statin — Statin Group: Conventional chemotherapy and maintenance therapy combined with statins.
  Arms: Statin Group
Drug: Sugar pill — Control Group: Conventional chemotherapy and maintenance therapy alone.
  Arms: Control Group

SUMMARY:
This study aims to evaluate the effect of statins combined with conventional chemotherapy and maintenance therapy on the prognosis of ovarian cancer patients, exploring its potential to improve survival rates and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants must provide written informed consent before any trial procedures commence. The consent form must be documented and retained at the research center.
* Female patients aged 18 years and older.
* Patients diagnosed with ovarian cancer, fallopian tube cancer, or primary peritoneal cancer (collectively referred to as ovarian cancer) through open surgery, laparoscopic surgery, or core needle biopsy confirmed by pathology.
* Patients who will require neoadjuvant chemotherapy followed by direct surgery, or direct surgical chemotherapy.
* Liver Function:

  1. Total bilirubin ≤1.5 times the upper limit of normal (ULN) or direct bilirubin ≤1.0 times ULN;
  2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times ULN. In cases of liver metastases, AST and ALT must be ≤5 times ULN.
* Kidney Function: Serum creatinine ≤1.5 times ULN, or creatinine clearance rate ≥60 mL/min (calculated using the Cockcroft-Gault formula).
* Participants must be able to understand the trial procedures and be capable of adhering to the trial protocol for the duration of the study. This includes the ability to complete any required treatments, examinations, tests, follow-up appointments, and questionnaires associated with the trial.

Exclusion Criteria:

* Are using other investigational drugs or participating in other clinical drug trials simultaneously;
* Have used or are currently using any medications that interact with statins;
* Have active cirrhosis, uncontrolled concurrent diseases, a history of chronic myopathy, active hepatitis, or unexplained persistent elevation of serum aminotransferases;
* Are known to be allergic to statins, or any active or inactive components of drugs with similar chemical structures;
* Are unable to swallow oral medications or have any gastrointestinal disorders that might interfere with the absorption and metabolism of the study drugs, such as uncontrolled nausea and vomiting, gastrointestinal obstruction, or malabsorption;
* Require treatment for symptomatic or uncontrolled brain metastases, including but not limited to surgery, radiation, and/or corticosteroids, or have clinical signs of spinal cord compression;
* Have severe, uncontrolled diseases or conditions that, in the investigator's judgment, make the participant unsuitable for the study. These include but are not limited to:

  1. Active viral infections such as HIV, hepatitis B, or hepatitis C.
  2. Severe cardiovascular diseases, including uncontrolled ventricular arrhythmias or a recent (within the last 3 months) myocardial infarction.
  3. Uncontrolled grand mal seizures, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorders affecting the ability to provide informed consent.
  4. Uncontrolled hypertension not managed by medication. Immune deficiencies (excluding splenectomy) or other conditions deemed by the investigator to pose a high risk of toxicity.
* Have any medical history or existing clinical evidence indicating the potential to confound study results, interfere with adherence to the trial protocol throughout the study, or not align with the patient's best interests;
* Have a history of or current evidence of other malignancies;
* Are pregnant, breastfeeding, or planning to become pregnant during the study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 12-month
  The time between the start of the trial and tumor progression (in any way) or death (from any cause)
Disease free survival | 12-month
  Time from surgical resection to local recurrence

SECONDARY OUTCOMES:
Changes of tumor marker CA125 | 12-month
  Changes in Serum CA125 from Enrollment to End of Trial
Changes of tumor marker HE4 | 12-month
  Changes in Serum HE4 from Enrollment to End of Trial
Lipid change | 12-month
  Changes in Serum Lipid from Enrollment to End of Trial

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Cancer Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No